CLINICAL TRIAL: NCT01746368
Title: Enabling Advance Directive Completion by Rural Alabama Veterans: A Pilot Study
Brief Title: Enabling Advance Directive Completion
Acronym: EADCRAV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: NRI 10-311
Record Dates: First submitted 2012-11-29; First posted 2012-12-10 (Estimated); Results first posted 2015-06-12 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-05

CONDITIONS: Advance Directives
Keywords: advance directives
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nurse-Supported Advance Care Planning Intervention (Experimental): The Nurse-Supported Advance Care Planning Intervention was a manualized education, support, and guidance session provided by a Registered Nurse that included information about risks, benefits, and alternatives of specific choices.
  Interventions: Other: The Nurse-Supported Advance Care Planning Intervention
- Care-as-Usual (Active Comparator): The Care-as-Usual was a session with the social worker who explained what the Advance Directive is, and guided the Veteran regarding the process of completing the Advance Directive document, without providing information about risks, benefits, and alternatives of specific choices. Subjects in this arm who desired information about risks, benefits, and alternatives of specific choices before randomization were scheduled for the Care-as-Usual session after they received that information from the Primary Care Provider.
  Interventions: Other: Care-as-Usual

INTERVENTIONS:
Other: The Nurse-Supported Advance Care Planning Intervention — This intervention was a manualized education, support, and guidance session provided by a Registered Nurse that included information about risks, benefits, and alternatives of specific choices. It incorporated an application of the Theory for Enabling Safety.
  Other Names: Enabling Intervention, RN session
  Arms: Nurse-Supported Advance Care Planning Intervention
Other: Care-as-Usual — The Care-as-Usual was a session with the social worker who explained what the Advance Directive is, and guided the Veteran regarding the process of completing the Advance Directive document, without providing information about risks, benefits, and alternatives of specific choices.
  Other Names: As Usual (AU) Intervention, SW session
  Arms: Care-as-Usual

SUMMARY:
Objectives: The objectives of the pilot study were to (1) test the feasibility of recruitment, randomization, and retention; (2) test the feasibility of a standardized Nurse-Supported Advance Care Planning Intervention; (3) evaluate the feasibility of the assessment process and data collection procedures; (4) evaluate the Veterans' satisfaction with the intervention and their Advance Directive decisions; and (5) evaluate preliminary effects of the Nurse-Supported Advance Care Planning Intervention.

Research Design: This was a prospective, randomized, controlled, unblinded pilot study. Alabama Veterans who received care through the Tuscaloosa VA Medical Center were randomized to either the Nurse-Supported Advance Care Planning Intervention or Care-as-Usual in a 2:1 ratio respectively. Data related to recruitment, randomization, and retention; study completion by subjects; completeness of data collection; Veterans' satisfaction; and preliminary effects of the intervention were collected, analyzed, and evaluated. The length of the study was one year.

Methods: The setting for the study was Tuscaloosa VA Medical Center care sites. A convenience sample of fifty subjects was recruited from Tuscaloosa VA outpatient clinics including Selma, residential settings, Home Based Primary Care, and the Mobile Health Unit. The level of care of subjects was all-inclusive, excepting current Hospice or Palliative Care. Selection procedures included self-referral and referral by Tuscaloosa VA Medical Center staff. Entry requirements were the meeting of all inclusion criteria and verification of no exclusion criteria. The Nurse-Supported Advance Care Planning Intervention was a manualized education, support, and guidance session provided by a Registered Nurse that included information about risks, benefits, and alternatives of specific choices. The Care-as-Usual was a session with the social worker who explained what the Advance Directive is, and guided the Veteran regarding the process of completing the Advance Directive document, without providing information about risks, benefits, and alternatives of specific choices. Study enrollment period was six months. The primary study outcome measure was Advance Directive completion rate. This pilot was not a hypothesis testing study. The underlying hypothesis of the eventual full study is that the Nurse-Supported Advance Care Planning Intervention is associated with Advance Directive completion rates at least comparable to that of the As-Usual care.

Significance: This study supports the Veterans Health Administration (VHA) mission to provide Veteran-centered care. It provides important information needed to plan a full study of the effectiveness of a specific Nurse-Supported Advance Care Planning Intervention to facilitate Advance Directive completion by rural Alabama Veterans.

DETAILED DESCRIPTION:
Background:

The VHA mission to serve the health care needs of America's veterans assumes a veteran-centered approach - one that evolves not only from the health team's assessment of needs, but especially one that begins with the veteran's assessment of his or her own needs. Preliminary data from the Alabama Veterans Rural Health Initiative study suggest that approximately 30% of rural Alabama veterans do not have an Advance Directive and want help completing one. Rural Alabama veterans live in counties with a higher percent of African American minorities, lower levels of education, and higher family poverty rates, than the average for the US population at large. Prior studies have demonstrated that disparities in Advance Directive completion rates may be related to race, level of income, and level of education. VHA research priorities include addressing the challenges of minority health care needs and the disparities that arise in healthcare delivery. Although many studies evidence the effectiveness of education and counseling in facilitating Advance Directive completion, data are lacking that demonstrate the efficacy of resource-conservative nursing interventions to enable Advance Directive completion by rural, southern minorities. This pilot lays the groundwork to address this evidence gap.

Objectives:

The objectives of the pilot study were to (1) test the feasibility of recruitment, randomization, and retention; (2) test the feasibility of a standardized Nurse-Supported Advance Care Planning Intervention; (3) evaluate the feasibility of the assessment process and data collection procedures; (4) evaluate the Veterans' satisfaction with the intervention and their Advance Directive decisions; and (5) evaluate preliminary effects of the Nurse-Supported Advance Care Planning Intervention.

Methods:

A prospective, randomized, controlled pilot study. Fifty Alabama veterans who receive care at the Tuscaloosa VA Medical Center were randomized to either the Nurse-Supported Advance Care Planning Intervention or Care-as-Usual. The Nurse-Supported Advance Care Planning Intervention was a manualized education, support, and guidance session provided by a Registered Nurse that included information about risks, benefits, and alternatives of specific choices. The Care-as-Usual was a session with the social worker who explained what the Advance Directive is, and guided the Veteran regarding the process of completing the Advance Directive document, without providing information about risks, benefits, and alternatives of specific choices. Data related to recruitment, randomization, and retention; study completion by subjects; completeness of data collection; Veterans' satisfaction; and preliminary effects of the intervention were collected, analyzed, and evaluated.

Status:

The Tuscaloosa VA Medical Center Institutional Review Board (IRB) has approved this study. Study is closed.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Male or female
* Any race or ethnic origin
* 19 years of age (i.e. minors are excluded)
* Veteran indicates he/she has no Advance Directive
* Speaks and understands English
* Any category of rurality through urbanity of home residence or place of habitation
* Veteran is willing to extend the screening/baseline visit or return within 30 days for the advance care planning (ACP) session

Exclusion Criteria:

* Diagnosis of dementia (all causes) or other cognitive disorder documented in computerized patient record system problem list. (Note: this would include, for example, a mental disability that precludes informed consent capacity, e.g. a documented condition including an age level equivalency understanding of a child of age 6)
* Diagnosis of serious mental illness (i.e. schizophrenia, schizoaffective disorder, bipolar I, major depression with psychotic features) documented in computerized patient record system problem list
* Actively considering plans of suicide or homicide per self report during screening interview direct question
* Psychotic symptoms that impair the subject's ability to give informed consent
* Current hospice care or palliative care recipient. (Note: The major predicted potential impact of this intervention is for Veterans who typically receive little or no ACP support. Veterans who receive palliative care/hospice care at Tuscaloosa VA Medical Center (VAMC) typically receive timely and full ACP support including Advance Directive completion support if desired. Veterans receiving palliative care and hospice care at Tuscaloosa VA Medical Center may tire easily and/or have pain/discomfort problems that could easily be exacerbated by research procedures. These research procedures themselves have the potential to add to end of life distress.)
* Currently incarcerated

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann F Mahaney-Price, BSN MS DNP, Principal Investigator — VA Medical Center, Tuscaloosa, AL
Locations (1):
- Tuscaloosa VA Medical Center, Tuscaloosa, AL, Tuscaloosa, Alabama, United States

REFERENCES:
- [Result] Ohlen J, Andershed B, Berg C, Frid I, Palm CA, Ternestedt BM, Segesten K. Relatives in end-of-life care--part 2: a theory for enabling safety. J Clin Nurs. 2007 Feb;16(2):382-90. doi: 10.1111/j.1365-2702.2006.01474.x. PMID 17239074

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From May 2013 - September 2013, 50 subjects were recruited from outpatient clinics, rural mobile clinic, home-based primary care, and residential treatment units.
Groups:
- Nurse-Supported Advance Care Planning Intervention: The Nurse-Supported Advance Care Planning Intervention was a manualized education, support, and guidance session provided by a Registered Nurse that included information about risks, benefits, and alternatives of specific choices. It incorporated an application of the Theory for Enabling Safety.
Period: Overall Study
Arm/Group | Nurse-Supported Advance Care Planning Intervention | Care-as-Usual
Started | 33 | 17
Recieved Allocated Intervention | 31 | 8
Assessment Completed | 31 | 16
Analyzed for AD Completion Rate | 32 | 17
Analyzed for Satisfaction | 30 | 16
Completed | 31 | 16
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: The number of participants for analysis was 50 - the full sample size.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nurse-Supported Advance Care Planning Intervention | Care-as-Usual | Total
Number analyzed (Participants) | 33 | 17 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 16 | 47
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.24 (11.48) | 48.35 (14.95) | 50.26 (12.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 26 | 15 | 41
Race/Ethnicity, Customized [Number; unit: Participants]
  White Non-Hispanic | 8 | 5 | 13
  Black Non-Hispanic | 21 | 9 | 30
  Black Hispanic | 0 | 1 | 1
  2 or more races Non-Hispanic | 3 | 1 | 4
  Other Non-Hispanic | 0 | 1 | 1
  Unknown/Not Reported | 1 | 0 | 1
Rurality [Number; unit: Participants]
  Rural zip code | 14 | 6 | 20
  Non-rural zip code | 19 | 11 | 30
Desire for Information About Advance Directives [Number; unit: Participants]
  Yes | 29 | 14 | 43
  No | 4 | 3 | 7
Desire for Help Completing an Advance Directive [Number; unit: Participants]
  Yes | 29 | 12 | 41
  No | 3 | 5 | 8
  No answer | 1 | 0 | 1
Desire for Risks, Benefits, and Alternatives Information About Life-sustaining Procedures [Number; unit: Participants]
  Yes | 29 | 10 | 39
  No | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed an Advance Directive
Description: An advance directive was considered completed upon confirmation of the scanned document in the medical record.
Time Frame: Up to 1 month after intervention
Population: intention to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Nurse-Supported Advance Care Planning Intervention | Care-as-Usual
Number analyzed (Participants) | 32 | 17
participants | 30 | 5

2. Secondary Outcome: Satisfaction
Description: Score on the Client Satisfaction Questionnaire-8 (CSQ-8). The overall score is produced by summing all item responses. For the CSQ-8, scores range from 8 to 32, with higher values indicating higher satisfaction.
  Response options differ from item to item, but all are based on a four-point scale.
  All items are positively worded; however, the directionality of response options span the spectrum from very negative to very positive; and, the numerical anchors for items are reversed randomly (from high to low or low to high) from item to item to minimize stereotypic response sets. The CSQ-8 has no subscales and reports a single score measuring a single dimension of overall satisfaction.
Time Frame: For participants who received the allocated intervention, up to one month after intervention; for all others, up to 90 days after consenting to the study.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Nurse-Supported Advance Care Planning Intervention | Care-as-Usual
Number analyzed (Participants) | 30 | 16
Scores on a scale | 31.03 (1.38) | 28.00 (4.13)

ADVERSE EVENTS:
Time Frame: Participants were followed for the duration of their participation in the study, up to 90 days.
Arm/Group | Nurse-Supported Advance Care Planning Intervention | Care-as-Usual
Serious Adverse Events (participants affected / at risk) | 1/33 | 1/17
Other Adverse Events (participants affected / at risk) | 1/33 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nurse-Supported Advance Care Planning Intervention (N=33) | Care-as-Usual (N=17)
Admission to acute psychiatric unit (Psychiatric disorders) | 1 (1) | 0 (0)
Admission to hospital (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nurse-Supported Advance Care Planning Intervention (N=33) | Care-as-Usual (N=17)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The local Institutional Review Board directed that the advance directive completion and satisfaction data for one participant randomized to the Nurse-Supported Advance Care Planning Intervention be excluded from analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No